CLINICAL TRIAL: NCT01447147
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Safety and Efficacy of CCX140-B in Diabetic Nephropathy
Brief Title: A Study to Evaluate the Safety and Efficacy of CCX140-B in Subjects With Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL005_140
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Nephropathy; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — CCX140-B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Group A) (Placebo Comparator)
  Interventions: Drug: Placebo
- CCX140-B (Group B) (Experimental)
  Interventions: Drug: CCX140-B
- CCX140-B (Group C) (Experimental)
  Interventions: Drug: CCX140-B

INTERVENTIONS:
Drug: Placebo — Placebo capsules once daily
  Arms: Placebo (Group A)
Drug: CCX140-B — CCX140-B capsules once daily (Group B)
  Arms: CCX140-B (Group B)
Drug: CCX140-B — CCX140-B capsules once daily (Group C)
  Arms: CCX140-B (Group C)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of treatment with CCX140-B in subjects with diabetic nephropathy.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of CCX140-B in subjects with diabetic nephropathy based on subject incidence of adverse events.

The secondary objectives of this study include evaluation of the effect of CCX140-B on several measures of effectiveness commonly used in the evaluation of diabetes and renal medications.

Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged 18-75 years inclusive, with documented previously diagnosed type 2 diabetes mellitus (per American Diabetes Association [ADA] criteria)
* Residual albuminuria despite stable treatment with an angiotensin-converting enzyme (ACE) inhibitor or an angiotensin receptor blocker (ARB) for at least 8 weeks prior to screening (Albumin:creatinine ratio [ACR] of 100 to 3000 mg/g creatinine, inclusive)
* Estimated glomerular filtration rate based on serum creatinine (eGFR, determined by Modification of Diet in Renal Disease [MDRD] equation) of ≥ 25 mL/min/1.73 m(2)
* Must be on a stable dose of an ACE inhibitor or ARB for at least 8 weeks prior to screening, but subjects must not be on both an ACE inhibitor and an ARB
* Hemoglobin A1c (HbA1c) > 6.0% but not > 10.0% and fasting plasma glucose less than 270 mg/dL at screening

Key Exclusion Criteria:

* Type 1 diabetes mellitus or history of diabetic ketoacidosis
* Previous renal transplant or known non-diabetic renal disease, except related to hypertension
* Undergone renal dialysis at any time in the past
* Received chronic (more than 7 days continuously) systemic glucocorticoid or other immunosuppressive treatment within 8 weeks of screening
* Use of bardoxolone, atrasentan or other endothelin antagonist within 8 weeks of screening
* Received chronic (more than 7 days continuously) non-steroidal anti-inflammatory drug (NSAID) treatment within 2 weeks of screening
* Cardiac failure (class III or IV), history of unstable angina, symptomatic coronary artery disease, myocardial infarction or stroke within 12 weeks of screening
* Poorly-controlled blood pressure (systolic blood pressure >155 or diastolic blood pressure >95, with blood pressure measured in the seated position after at least 5 minutes of rest)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2011-10; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Subject incidence of adverse events | Up to 365 days
  The primary objective of this study is to evaluate the safety and tolerability of CCX140-B in subjects with diabetic nephropathy.

SECONDARY OUTCOMES:
Change from baseline in first morning urinary albumin:creatinine ratio (ACR) | Up to 365 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (83):
- Belgium (7):
  - Antwerp
  - Brussels
  - Edegem
  - Ghent
  - Leuven
  - Liège
  - Roeselare
- Czechia (14):
  - Beroun
  - Brno
  - Hlučín
  - Neratovice
  - Nový Jičín
  - NZdar Nad Sazavou
  - Pardubice
  - Prague
  - Přelouč
  - Rakovník
  - Slaný
  - Třebíč
  - Uherský Brod
  - Uničov
- Germany (18):
  - Berlin
  - Bosenheim
  - Cologne
  - Deggingen
  - Dresden
  - Erlangen
  - Hanover
  - Heidelberg
  - Heilbronn
  - Hoyerswerda
  - Munich
  - Neuwied
  - Nuremberg
  - Pirna
  - Potsdam
  - Saarlouis
  - Speyer
  - Wiesbaden
- Hungary (13):
  - Baja
  - Balatonfüred
  - Békéscsaba
  - Budapest
  - Debrecen
  - Eger
  - Gyula
  - Hatvan
  - Kaposvár
  - Kisvárda
  - Sátoraljaújhely
  - Szekszard, Tolna
  - Szikszó
- Poland (11):
  - Bialystok
  - Ciechanów
  - Gdansk
  - Grodzisk Mazowiecki
  - Krakow
  - Poznan
  - Radom
  - Rzeszów
  - Szczecin
  - Warsaw
  - Wroclaw
- United Kingdom (20):
  - Bath
  - Belfast
  - Birmingham
  - Bristol
  - Chester
  - Coventry
  - Doncaster
  - Edmonton
  - Liverpool
  - Livingston
  - London
  - Londonderry
  - Manchester
  - Middlesbrough
  - Norfolk
  - Preston
  - Salford
  - Sheffield
  - Swansea
  - Welwyn Garden City

REFERENCES:
- [Derived] de Zeeuw D, Bekker P, Henkel E, Hasslacher C, Gouni-Berthold I, Mehling H, Potarca A, Tesar V, Heerspink HJ, Schall TJ; CCX140-B Diabetic Nephropathy Study Group. The effect of CCR2 inhibitor CCX140-B on residual albuminuria in patients with type 2 diabetes and nephropathy: a randomised trial. Lancet Diabetes Endocrinol. 2015 Sep;3(9):687-96. doi: 10.1016/S2213-8587(15)00261-2. Epub 2015 Aug 9. PMID 26268910
- [Derived] Sullivan T, Miao Z, Dairaghi DJ, Krasinski A, Wang Y, Zhao BN, Baumgart T, Ertl LS, Pennell A, Seitz L, Powers J, Zhao R, Ungashe S, Wei Z, Boring L, Tsou CL, Charo I, Berahovich RD, Schall TJ, Jaen JC. CCR2 antagonist CCX140-B provides renal and glycemic benefits in diabetic transgenic human CCR2 knockin mice. Am J Physiol Renal Physiol. 2013 Nov 1;305(9):F1288-97. doi: 10.1152/ajprenal.00316.2013. Epub 2013 Aug 28. PMID 23986513